CLINICAL TRIAL: NCT06649227
Title: Prospective Non-randomized Phase I Study Investigating the Safety of CD19 CAR-T Cells in Patients With Refractory/Relapsed AML Expressing CD19.
Brief Title: Study Investigating the Safety of CD19 CAR-T Cells in Relapsed/Refractory AML Expressing CD19
Acronym: CARLA-M19
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government); University Hospital, Rouen (Other); Miltenyi (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021_0578; 2023-509212-29-01 (EU CTIS Number)
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Relapsed Adult AML
Keywords: Relapsed/refractory AML expressing CD19; AML; CD19; CAR-T cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Other)
  Interventions: Drug: CAR-T cell therapy

INTERVENTIONS:
Drug: CAR-T cell therapy — cyclophosphamide and fludarabin conditioning , followed by a target dose of 1 x 10exp6 of autologous, genetically modified, anti-CD19 CAR-T cells per kg of body weight.

SUMMARY:
Refractory/Relapsed (R/R) acute myeloid leukemia (AML) is associated with a dis-mal prognosis.

In some subsets of AML such as AML driven by the t(8;21) translocation, leading to the RUNX1-RUNX1T1 (AML1-ETO) fusion transcript expression, CD19 B-cell antigen is aberrantly expressed on malignant blasts in around 80 % of cases. Interestingly, the expression of the CD19 antigen is also detected in the CD34+ CD38-population leukemic stem cells.

t(8;21) AML subtype has a rather good prognosis with an intensive chemotherapy regimen, but relapses occur in around 40 % of the patients and new therapeutic options are needed for these patients.

Plesa et al, reported a successful treatment of a refractory t(8;21) AML with bispecific monoclonal antibodies that targets CD19. More recently, Danylesko et al, have reported long-term remission following CD19 CAR-T cells in a heavily pre-treated patient with t(8;21) AML(1). The same group has just submitted an abstract of 6 treated patients to the European Haematology Association (EHA) 2023 meet-ing: Six patients (adults-5, child-1) with t(8; 21) AML (confirmed by cytogenetic and FISH) and aberrant CD19 expression were included. One patient had a complex karyotype. Molecular analysis for CKIT, NPM1, IDH1, IDH2, and CBPa were nega-tive in all pts. One pt harbors the FLT3 ITD and TKD mutations. Median number of previous chemotherapy (CT) lines was 4 (3-8). Four patients were with chemo re-sistant relapse post allo-HCT (MSD-1, 10/10 MUD -3) 5-18 months before CAR T-cell infusion. All patients developed CRS (grade 1-3) and were treated with i.v tocili-zumab and dexamethasone. 2/6 patients suffered from ICANS and were treated with steroids. In 4/6 patients, day 28 BM aspiration disclosed normal hematopoie-sis with no excess blasts and lack of t(8;21) by FISH confirming clinical and cyto-genetic remission, while 2/6 pts with progressive AML had no response (Danylesko etal. Abstract EHA 2023, submitted).

Interestingly, other subsets of AML display an aberrant expression of CD19. These observations indicate that CD19 can be a target of choice for CAR-T cells in patients with R/R AML expressing this antigen.

In this study, we plan to offer anti-CD19 CAR-T cell therapy to patients with re-lapsed/refractory AML expressing CD19 for whom no curative alternatives are available.

To this end, CAR-T cells will be manufactured using closed semi-automated bioreactor CliniMACS Prodigy (Miltenyi Biotec) in academic setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age at the time of signing the informed consent form,
* Patient with AML that expresses CD19 by Flow-cytometry, (CD19 expression ≥ 70% of AML blasts)
* Patients with R/R AML defined as:

  * Primary refractory: absence of remission after two courses of induction chemotherapy,
  * Secondary refractory: absence of remission after salvage treatment in relapsing patients,
  * Post-transplant relapse in patients having had allo-HCT.
* Lack of accessible targeted therapy that has not been previously utilized.
* Eastern Cooperative Oncology Group (ECOG) performance status of < 2,
* Estimated life expectancy of > 2 months,
* Magnetic resonance imaging (MRI) of the brain showing no evidence of central nervous system (CNS) involvement,
* Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1 (except for clinically non-significant toxicities, such as alopecia),
* Platelet count ≥ 30000/uL,
* Absolute lymphocyte count ≥ 200/uL,
* Creatinine clearance (as estimated by Cockcroft Gault) ≥ 40 mL/min,
* Serum ALT/AST ≤ 2.5 upper limit of normal (ULN),
* Total bilirubin ≤ 1.5 mg/dl, except in subjects with Gilbert's syndrome,
* Cardiac ejection fraction ≥ 45 %,
* No clinically significant electrocardiogram (ECG) findings,
* No clinically significant pleural effusion,
* Baseline oxygen saturation > 92 % on room air,
* Female patients of childbearing potential must:

  1. have a negative pregnancy test (blood) at screening visit.
  2. either commit to true abstinence from heterosexual contact or agree to use, and be able to comply with, effective measures of contraception without interruption, from screening through 1 year following the CAR-T cell infusion. A highly effective method of contraception or birth control (failure rate less than 1% per year when used consistently and correctly) must be practiced. The patient should be informed of the potential risks associated with becoming pregnant while enrolled in this clinical trial. Reliable methods for this trial are: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, sexual abstinence or vasectomized sexual partner. Abstinence is only accepted as true abstinence: when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods and withdrawal] are not acceptable methods of contraception.) Postmenopausal (no menses for at least 1 year without alternative medical cause) or surgically sterile female patients (tubal ligation, hysterectomy or bilateral oophorectomy) may be enrolled.
  3. Agree to abstain from breast feeding during the study participation and for 1 year after the CAR-T cell infusion.
* Male patients must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential for at least 1 year after the CAR-T cell infusion, even if he has undergone a successful vasectomy.

Exclusion Criteria:

* Patient unable to sign the informed consent,
* Patient with R/R AML that does not expresses CD19,
* History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) unless disease-free and without anticancer therapy for at least 3 years,
* Prior CD19 targeted therapy,
* Prior CAR therapy or other genetically modified T cell therapy,
* Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management,
* History of human immunodeficiency virus (HIV) or HTLV1,
* Infection or acute or chronic active hepatitis C infection,
* Infection or acute or chronic active hepatitis (Hep) B. Subjects with history of Hep B or Hep C infection must have cleared their infection as determined by standard serological and genetic testing per current Infectious Diseases Society of America (IDSA) guidelines,
* Subjects with detectable cerebrospinal fluid malignant cells or known brain metastases or with a history of cerebrospinal fluid (CSF) malignant cells or brain metastases,
* History or presence of non-malignant CNS disorder, such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement,
* Patient placed under guardianship or curatorship,
* Females either pregnant/breast-feeding or planning to become pregnant,
* Any contraindication due to hypersensitivity to the active substance or to any of the excipients,
* Contraindication to the lymphodepleting chemotherapy,
* Absence of medical insurance cover.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2029-07-10 (Estimated); Study Completion 2030-07-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients deceased without progression one month after CAR-T cell infusion | at 1 month
  Non-progression mortality (NPM), type and frequency of adverse events. NPM is defined as death occurred in patients without evidence of AML progression. Absence of response, progression or relapse of AML define progression status

SECONDARY OUTCOMES:
Number of patients with manufacturing failure and out of specification (OOS) deviation | Througth study completion, an average of 2 years
Duration of CAR-T cell persistence in blood after infusion evaluated by flow-cytometry and PCR, | Througth study completionan, average of 2 years
Number of patients with overall response | at 1 month
Response duration | at 3 months, 6 months and 12 months
Number of patients alive | at 3 months, 6 months and 12 months
Number of patients alive without relapse | at 3 months, 6 months and 12 months
Number of deaths without progression | at 3 months, 6 months and 12 months
Number of patients with complete remission (CR) | at 1 month and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Yakoub-Agha, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No